CLINICAL TRIAL: NCT04868643
Title: A Prospective Multicenter, Open Label, Non-Randomized, Cross-Over Study Evaluating the Use of the DIMI Renal Replacement Therapy (RRT) System In-Center by Trained Dialysis Nurses and In-Home by Trained Care Partners and Patients With End Stage Renal Disease (ESRD) Who Are on Stable Dialysis Regimens.
Brief Title: The Evaluation of the DIMI RRT System In-Center to Demonstrate Safety and Usability in the Home Environment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The company no longer wishes to pursue this IDE
Sponsor: Dialco Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIAL-DIMI-001
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: ESRD; Hemodialysis
Keywords: Home Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Replacement Therapy; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- In-Center arm (Other): Subjects undergo In-Center treatment in Phase 2 as defined.
  Interventions: Device: The DIMI Renal Replacement Therapy (RRT) System
- In-Home arm (Other): Subjects undergo In-Home treatments in Phase 4 as defined.
  Subjects in Phase 2 and Phase 4 will be the same.
  Interventions: Device: The DIMI Renal Replacement Therapy (RRT) System

INTERVENTIONS:
Device: The DIMI Renal Replacement Therapy (RRT) System — To demonstrate that the safety and efficacy of the DIMI RRT remains consistent when used In-Center by trained dialysis nurses versus in an In-Home environment by trained Care Partners and Subjects.

SUMMARY:
This is a prospective, multicenter, open label, non-randomized, cross-over study. Subjects will be enrolled in the trial for approximately 18 weeks and will use the DIMI RRT System for their dialysis treatments for all study phases, according to the schedule outlined below. The schedule will consist of four phases and the number of sessions per week will be prescribed the same throughout Phase 1 to 4.

DETAILED DESCRIPTION:
1. Phase 1: Run-in. Duration: 2 weeks. Potential Subjects will undergo dialysis treatments 3 - 5 times per week for up to 2 weeks In-Center. Treatments will be administered by study staff during this phase. Study eligibility will be assessed for both the potential Subject and their Care Partner after completion of the run-in period. Potential subjects and Care Partners who meet all eligibility criteria will be invited to Phase 2.
2. Phase 2: In-Center Treatment. Duration: 6 weeks. Subjects will undergo dialysis treatments 3 - 5 times per week for approximately 6 weeks (for a total of 18 - 30 sessions) In-Center. Treatments will be administered by study staff.
3. Phase 3: Cross-over Period from In-Center to In-Home environment. Duration: 4 weeks. Care Partners will undergo the DIMI training, then perform dialysis treatments on Subjects 3 - 5 times per week for approximately 4 weeks (for a total of 12 - 20 sessions). Treatments will be completed In-Center under the supervision of hemodialysis nurses and at the discretion of the investigator.
4. Phase 4: In-Home Treatment. Duration: 6 weeks. Care Partners will perform dialysis treatments to the Subject 3 - 5 times per week for approximately 6 weeks (for a total of 18 - 30 sessions) in a home environment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent and has signed a Health Insurance Portability and Accountability Act of 1996 (HIPAA) compliant authorization statement.
2. Subject is at least 18 years and less than 75 years of age.
3. Subject has identified an individual "Care Partner" to be trained and available as needed. Such Care Partner must be considered competent to train on the use of the device by the prescribing physician, and must commit to the trial.
4. Subject has end stage renal disease (ESRD) adequately treated by maintenance dialysis achieving a Kt/V ≥ 1.2 and has been deemed stable for at least three months by his/her treating nephrologist.
5. Subject has a well-functioning and stable vascular access that allows a blood flow of at least 300 ml/min.
6. Subject has a documented psychosocial evaluation by a qualified social worker, treating physician or home hemodialysis nurse.
7. Subject has no childbearing potential or has a negative pregnancy test within 7 days prior to the start of the first study treatment and will be utilizing medically acceptable means of contraception during the study period.
8. Subject has a home environment to perform hemodialysis that meets the criteria of Home Use Environment (defined in Section 15.1).

Exclusion Criteria:

1. Subject has dementia or lacks capacity for self-care.
2. Life expectancy less than 12 months from first study procedure.
3. Subject is unable to understand or cooperate with hemodialysis nurse and dialysis care team.
4. Subject has a documented history of non-adherence to dialysis treatment that would prevent successful completion of the study.
5. Subject has had a recent major cardiovascular adverse event within the last 3 months.
6. Subject has New York Class III or IV Congestive Heart Failure, or ejection fraction less than 30%.
7. Subject has a persistent pre-dialysis sitting systolic blood pressure less than 100 mmHg despite medical therapy.
8. Subject has symptomatic intra-dialytic hypotension requiring medical intervention in two of their last three treatments.
9. Subject has an active infection requiring antibiotics within the last 7 days.
10. Subject has fluid overload due to intractable ascites secondary to liver cirrhosis.
11. Subject has uncontrolled blood pressure (e.g. sustained/persistent pre- dialysis systolic blood pressure greater than 180 mmHg despite maximal medical therapy in two of the last three treatments).
12. Subject is intolerant to heparin.
13. Subject is seroreactive for Hepatitis B Surface Antigen.
14. Subject has an active, life-threatening, rheumatologic disease.
15. Subject has a history of adverse reactions to dialyzer membrane material.
16. Subject is participating in another investigative drug or device clinical study related to Home Hemodialysis which conflicts with the execution of this study.
17. Subject is expected to receive a kidney transplant from any donor organ in the next 6 months.
18. Subject has a life-threatening malignancy actively receiving treatment that would prevent successful completion of the study protocol.
19. Any other condition that the Investigator feels would prevent the Subject from being a suitable candidate for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Delivery of the prescribed fluid volume, defined as delivered volume that is at least 90% of prescribed volume at each in-home dialysis session. | 6 weeks
  The delivered volume is the total effluent volume (spent dialysate plus net ultrafiltrate) as measured by the device by means of 2 independent and calibrated electronic scales. The effluent volume is an effective means of assessing the usability of the machine in different environments and by different people, as any early interruption of treatment will result in a lower delivered volume.

SECONDARY OUTCOMES:
Delivery of a standardized weekly Kt/V based on lab data. | 6 weeks
  The secondary efficacy endpoint is the delivery of a standardized weekly Kt/V of greater than or equal to 2.1, that will be measured weekly. The standardized weekly Kt/V value will be computed by the Sponsor and included in the study database from laboratory data provided and recorded by the site via the Case Report Forms (CRFs).

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan for IPD sharing